CLINICAL TRIAL: NCT00823914
Title: Developing A Validated Measure of the Impact of Psoriasis on Chronic Quality of Life
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexandra Kimball, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2008P002090
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Quality of Life
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective of the study is to create and validate Chronic Quality of Life (CQOL) index that explores habits, career paths and other life choices psoriasis patients make as a result of coping with their disease that may not be impacted by therapy implemented at a given point in time.

- The investigators think this data will show that patients who were diagnosed at a young age will have worse chronic quality of life.

DETAILED DESCRIPTION:
As a visible disease, psoriasis can be embarrassing and psychosocially stressful in addition to physically uncomfortable. Patients' lives are affected in physical, psychological, social, sexual and occupational aspects. These burdens may cause patients to assume maladaptive habits and coping mechanisms, leading to a downward spiral in functioning within society, prohibiting patients from achieving their highest potential quality of life.

The investigators' study goal is to create and validate Chronic Quality of Life (CQOL) index that explores habits, career paths and other life choices psoriasis patients make as a result of coping with their disease that may not be impacted by therapy implemented at a given point in time. In creating this questionnaire and validating it the investigators will collect preliminary data. The investigators think this data will show that patients who were diagnosed at a young age will have worse chronic quality of life. In the long run, the investigators will use the CQOL index in studies in which patients are treated for psoriasis to determine which treatments can change a psoriasis patient's chronic quality of life. This information will be used to create guidelines for treatment focused on achieving a patient's optimal quality of life.

Another aspect that the investigators would like to look at is the skin carotenoid levels in the psoriasis population. Previous studies showed that psoriasis patients had lower levels of skin carotenoids when compared to healthy volunteers. This observation was not statistically significant perhaps due to a small sample size (21 subjects in the psoriasis group and 35 subjects in the control group). Skin carotenoid levels measurement is optional for study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent
* Able to read English
* Able to comply with study procedure
* Male or female of at least 18 years of age
* Has a diagnosis of psoriasis

Exclusion Criteria:

* Has any medical condition that might interfere with ability to complete CQOL survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psoriasis patients aged 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2008-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Chronic Quality of Life (CQOL) survey validation. | 1 year

SECONDARY OUTCOMES:
Skin carotenoid levels | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital CURTIS, Boston, Massachusetts, United States